CLINICAL TRIAL: NCT02557841
Title: Effects of Cerebellar Transcranial Direct Current Stimulation (ctDCS) on Motor Learning of Healthy Individuals
Brief Title: Cerebellar tDCS on Motor Learning of Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, PhD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Cerebellar_tDCS_MotorLearning
Record Dates: First submitted 2015-09-01; First posted 2015-09-23 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Cerebellum; Transcranial Direct Current Stimulation; Motor Learning; Serial Reaction Time Task; Handwriting
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- anodal ctDCS (Experimental): Volunteers will be submitted to anodal ctDCS + motor learning assessments (SRTT and Handwriting test).
  Interventions: Device: tDCS
- cathodal ctDCS (Experimental): Volunteers will be submitted to cathodal ctDCS + motor learning assessments (SRTT and Handwriting test).
  Interventions: Device: tDCS
- sham ctDCS (Sham Comparator): Volunteers will be submitted to sham ctDCS + motor learning assessments (SRTT and Handwriting test)
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Current will be applied by a DC stimulator (NeuroConn Plus, Germany).The active electrode (anode: 5x7 cm²) will be placed over the left cerebellar hemisphere (3 cm lateral to the inion) and the reference (5x7 cm²), over the left arm with current intensity of 2mA, fade in and fade out of 10 seconds, during 20 minutes.
  Arms: anodal ctDCS
Device: tDCS — Current will be applied by a DC stimulator (NeuroConn Plus, Germany). The active electrode (cathode: 5x7 cm²) will be placed over the left cerebellar hemisphere (3 cm lateral to the inion) and the reference (5x7 cm²), over the left arm with current intensity of 2mA, fade in and fade out of 10 seconds, during 20 minutes.
  Arms: cathodal ctDCS
Device: tDCS — Sham ctDCS (NeuroConn Plus, Germany) will be applied at the same parameter settings used on cathodal ctDCS however, current duration will be only 30 seconds. Moreover, device automatically turned off without volunteer's perception, but volunteers will be with electrodes montage for 20 minutes.
  Arms: sham ctDCS

SUMMARY:
A crossover trial with healthy volunteers will be conducted. Three sessions will be performed with at least 48 hours washout period to minimize carry-over effects. In each session, volunteers will be submitted to: fatigue and attention levels evaluation, handwriting test, serial reaction time task (SRTT) before and after ctDCS conditions and after session, a performance perception evaluation.

DETAILED DESCRIPTION:
A crossover, pseudo-randomized, sham-controlled and triple blind will be performed in order to evaluate ctDCS effects on motor learning, since evidence pointed to the crucial role of cerebellum on motor behavior. A non-involved research will conduct a pseudo-randomization (www.randomization.com) to warrant the counterbalanced sessions order and the allocation concealment. Volunteers, researchers and statistical analysis will be blinded to ctDCS condition.

After given prior informed consent, volunteers will be submitted to three experimental sessions: anodal ctDCS, cathodal ctDCS and sham ctDCS. Fatigue and attention levels, handwriting test and SRTT will be performed before and after stimulation. In addition, performance perception evaluation will be assessed at the end of session.

Electrical current will be delivered through a DC stimulator (NeuroConn Plus, Germany) using a pair of saline-soaked sponge electrodes (surface 35cm²). The active electrode (anode or cathode) will be placed over the left cerebellum (3 cm lateral to the inion) and the reference, over the left arm with current intensity of 2mA, fade in and fade out of 10 seconds, during 20 minutes. Sham tDCS has been used in several studies to evaluate active tDCS effects.

Sham ctDCS will be applied using the same electrodes placement and parameter settings of cathodal ctDCS however, stimulation will last only 30 seconds but volunteers will be with electrodes montage for 20 minutes. Because the device will be automatically turned off without volunteer's perception, early sensations (mild to moderate tingling) on stimulation site will be experienced without inducing any modulatory effects. Moreover, after each ctDCS session, an adverse effects questionnaire will be applied.

Fatigue and attention levels will be measured through an analogue scale graded from 0 to 10, where 0 means lower fatigue or attention levels and 10, the higher fatigue or attention levels.

Handwriting test: volunteers will be instructed to write six words with digital pen using the non-dominant hand on a tablet provided with analysis software system (MovAlyzer, EUA). The task will be performed spontaneously, without any instruction bias during writing activity. Each session has different word sequences but the difficulty level will be maintained (six words, two of them with 4, 6 and 8 letters).

SRTT: will be performed through software with visual stimuli presented on a computer screen in four different positions. Volunteer must press, with the non-dominant hand, a corresponding key with a predetermined finger as soon as possible when a highlighted star appears on the screen. The test comprises eight blocks with 120 trials each. Implicit motor learning is measured by performance changes between the blocks 5, 6 and 7.

Performance perception evaluation: in order to correlate stimulation type to the conscious improvement on motor task performance (SRTT and handwriting test) will be asked in the end of each session: "Regarding today's session, comparing your motor performance before and after cerebellar stimulation, you consider that you were better, worse or the same as before?"

ELIGIBILITY:
Inclusion Criteria:

* Right-handed (assessed by Edinburgh Handedness Inventory)
* Healthy volunteers (self report)
* Absence of neurological and psychiatric diseases
* No history of severe musculoskeletal injury on wrists and fingers
* Without using drugs or neuroactive substances regularly

Exclusion Criteria:

* Pregnancy
* Presence of metallic implant in close contact to the target stimulation area
* Acute eczema under the target stimulation area
* Pacemaker
* History of seizures or epilepsy
* Hemodynamic instability

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Changes on implicit motor learning | One week (before and after ctDCS)
  Serial reaction time task evaluates implicit motor learning through software with visual stimuli presented on a computer screen in four different positions. Volunteer must press, with the non-dominant hand, a corresponding key with predetermined fingers as soon as possible when a highlighted star appears on the screen. The test comprises eight blocks with 120 trials each.

SECONDARY OUTCOMES:
Changes on fatigue levels | One week (before and after ctDCS)
  It will be measured through an analogue scale graded from 0 to 10, where 0 means lower fatigue levels and 10, the higher fatigue levels.
Changes on attention levels | One week (before and after ctDCS)
  It will be measured through an analogue scale graded from 0 to 10, where 0 means lower attention levels and 10, the higher attention levels.
Changes on explicit motor learning | One week (before and after ctDCS)
  Handwriting test is an explicit motor learning measure. Volunteers will be instructed to write six words with digital pen using the non-dominant hand on a tablet provided with analysis software system (MovAlyzer, EUA). The task will be performed spontaneously, without any instruction bias during writing activity.

OTHER OUTCOMES:
Changes on performance perception | One week (after each session)
  in order to correlate stimulation type to the conscious improvement on motor task performance (SRTT and handwriting test) will be asked in the end of each session: "Regarding today's session, comparing your motor performance before and after cerebellar stimulation, you consider that you were better, worse or the same as before?"
Cerebellar tDCS adverse effects | One week (after each session)
  It will be evaluated through structured questionnaires that include most common stimulation sensations.

CONTACTS AND LOCATIONS:
Overall Officials: Kátia K Monte-Silva, PhD, Study Director — Universidade Federal de Pernambuco
Locations (1):
- Applied Neuroscience Laboratory, Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil